CLINICAL TRIAL: NCT05262283
Title: Has The COVID-19 Pandemic Affected Injury in Football? Example of a Professional Football Team
Brief Title: Has The COVID-19 Pandemic Affected Injury in Football?
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nurhayat KORKMAZ, Research assistant, Karadeniz Technical University
Other Study IDs: KTU-NK-TS-01
Record Dates: First submitted 2022-02-28; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Injuries
Keywords: COVID-19; Football; Injuries
MeSH Terms: conditions — Wounds and Injuries; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2019-2020 season: Injuries in the first 26 games of 2019-2020
  Interventions: Other: No intervention
- 2020-2021 season: Injuries in the first 26 games of 2020-2021 in the new post-COVID season
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention was made.

SUMMARY:
This study aims to compare the injuries that occurred in the football players after the isolation and lack of training caused by New Coronavirus Disease (COVID-19), with the previous season, based on the example of a professional football team in Turkey.

DETAILED DESCRIPTION:
This study aims to compare the injuries that occurred in the football players who faced an intense match tempo after the isolation and lack of training caused by COVID-19, as well as the stress and uncertainty, with the previous season, based on the example of a professional football team in Turkey. Injury follow-up data were examined.

ELIGIBILITY:
Inclusion Criteria:

* Having a musculoskeletal injury during the official match or team training in the 2019-2020 or 2020-2021 season

Exclusion Criteria:

* Signing a contract with Trabzonspor A Team in the 2020-2021 season

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants consist of professional football players who have a contract with the A team.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of injuries | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  The number of injuries in the two seasons was recorded separately.
Injury time | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Training injuries, Match injuries
Injury severity | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Minor, moderate, major
Injury type | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Sprain, strain, fracture, contision, other
Injury location | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Foot, ankle, calf, knee, thigh, hip, groin, lumbal
Injured tissue | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  muscle, tendon, tendon bone junction, capsule, ligament, bone, aponeurosis, meniscus
Injured side | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Left, right
Injury mechanism | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  noncontact, contact
Rule violation | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Opponent, no
Recurrence | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Yes, no

SECONDARY OUTCOMES:
Training | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  The number of days away from training
Missed Matches | Change of data in the first 26 matches of the 2019-2020 and 2020-2021 seasons
  Number of official matches missed

CONTACTS AND LOCATIONS:
Overall Officials: Nurhayat Korkmaz, PhDstudent, Principal Investigator — Karadeniz Technical University
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)